CLINICAL TRIAL: NCT01336010
Title: Treatment of Recently Acquired Hepatitis C Virus Infection
Acronym: ATAHC-II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R01DA015999-07 (NIH)
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Acute Hepatitis C
Keywords: Hepatitis C; Acute Hepatitis C; Early chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group A - 8 weeks therapy (Experimental): 8 weeks total of Pegylated interferon and ribavirin if undetectable HCV RNA after 2 weeks of therapy.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Group B - 16 weeks therapy (Experimental): 16 weeks total of Pegylated interferon and ribavirin if undetectable HCV RNA after 4 weeks of therapy.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Group C - 24 weeks therapy (Experimental): 24 weeks total of Pegylated interferon and ribavirin if undetectable HCV RNA after 6 weeks of therapy.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Group D - 32 weeks (gt1) or 24 weeks (gt 2/3) (Experimental): 32 weeks total of Pegylated interferon and ribavirin if undetectable HCV RNA after 8 weeks of therapy (genotype 1) or 24 weeks total of Pegylated interferon and ribavirin if undetectable HCV RNA after 8 weeks of therapy.
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Group E - 48 weeks (gt 1) or 24 weeks (gt 2/3) (Experimental): 48 weeks total of Pegylated interferon and ribavirin if undetectable HCV RNA after 12 weeks of therapy (genotype 1) or 24 weeks total of Pegylated interferon and ribavirin if undetectable HCV RNA after 12 weeks of therapy (genotype 2/3).
  Interventions: Drug: Peginterferon alfa-2a; Drug: Ribavirin
- Untreated Group (No Intervention): Observation only. No treatment for hepatitis C administered. Subjects who have undetectable HCV RNA at baseline, do not wish to commence treatment or are ineligible for treatment.

INTERVENTIONS:
Drug: Peginterferon alfa-2a — PEG-IFN 180 mcg in 0.5 ml (prefilled syringes) administered subcutaneously (SC) once weekly
  Other Names: Pegasys
  Arms: Group A - 8 weeks therapy; Group B - 16 weeks therapy; Group C - 24 weeks therapy; Group D - 32 weeks (gt1) or 24 weeks (gt 2/3); Group E - 48 weeks (gt 1) or 24 weeks (gt 2/3)
Drug: Ribavirin — Genotype 1: 1000mg or 1200mg p.o. daily in split doses (1000mg for patients weighing <75kg and 1200mg for patients weighing ≥ 75kg) Genotypes 2/3: 800mg daily p.o. daily in split doses for genotype 2 and 3 patients
  Arms: Group A - 8 weeks therapy; Group B - 16 weeks therapy; Group C - 24 weeks therapy; Group D - 32 weeks (gt1) or 24 weeks (gt 2/3); Group E - 48 weeks (gt 1) or 24 weeks (gt 2/3)

SUMMARY:
To determine whether response guided treatment with pegylated interferon +/- ribavirin is effective for the treatment of recently acquired hepatitis C infection. Response guided treatment is when the length of treatment is determined by how quickly you respond to the treatment.

DETAILED DESCRIPTION:
A prospective longitudinal study of natural history and treatment outcomes following response guided treatment of recent hepatitis C infection.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 16 years of age
* Recent hepatitis C infection with an estimated duration of Infection ≤ 18 months defined as

A)

* i) First anti-HCV antibody or HCV RNA positive within the previous 6 months and
* ii) Documented anti-HCV antibody negative or HCV RNA negative within the 24 months prior to anti-HCV antibody positive result

OR

B)

* i) First anti-HCV antibody or HCV RNA positive within the previous 6 months and
* ii) acute clinical hepatitis (jaundice or ALT> 10 X ULN) within the 12 months prior to first positive HCV antibody or HCV RNA with no other cause of acute hepatitis identifiable and
* Adequate English to provide written, informed consent and to provide reliable responses to the study interview
* Provision of written, informed consent.

Exclusion Criteria:

All patients:

• Individuals considered by the study investigators to be unlikely to participate in intensive follow-up and/or unwilling to provide extra blood samples

Treatment group only:

* Age between 16 and 18 years
* Women with ongoing pregnancy or breast feeding
* Therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) *6 months prior to the first dose of study drug
* Any investigational drug <6 weeks prior to the first dose of study drug
* Positive test at screening for anti-HAV IgM Ab, anti-HBc IgM Ab
* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g. hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease
* Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening
* Serum creatinine level >1.5 times the upper limit of normal at screening
* Hgb< 12g/dL in women or < 13g/dL in men at screening (for patients who receive combination therapy with PEG-IFN and ribavirin only)
* Male partners of women who are pregnant (for patients who receive combination therapy with PEG-IFN and ribavirin only)
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease
* Evidence of severe retinopathy (e.g. CMV retinitis, macular degeneration)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and efficacy of response-guided pegylated interferon and ribavirin for the treatment of recent HCV infection. Response-guided means the duration of treatment will be determined by the subject's early response to treatment. | 8-48 weeks
  Treatment duration will be determined by time to undetectable HCV RNA. Undetectable at week 2=8 weeks of therapy; Undetectable at week 4=16 weeks of therapy; Undetectable at week 6=24 weeks of therapy; Undetectable at week 8=32 weeks of therapy (24 weeks for genotypes 2/3); Undetectable at week 12=48 weeks of therapy (24 weeks for genotypes 2/3);

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Dore, MBBS, PhD, Principal Investigator — University of New South Wales
Locations (8):
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Kirketon Road Centre, Darlinghurst, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - St Vincent's Hospital Melbourne, Melbourne, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria

REFERENCES:
- [Derived] Martinello M, Hellard M, Shaw D, Petoumenos K, Applegate T, Grebely J, Yeung B, Maire L, Iser D, Lloyd A, Thompson A, Sasadeusz J, Haber P, Dore GJ, Matthews GV. Short duration response-guided treatment is effective for most individuals with recent hepatitis C infection: the ATAHC II and DARE-C I studies. Antivir Ther. 2016;21(5):425-34. doi: 10.3851/IMP3035. Epub 2016 Feb 11. PMID 26867206